CLINICAL TRIAL: NCT03454516
Title: Mobility Hypertension Management - Effect of Telemonitoring on Hypertension Management
Brief Title: Mobility Hypertension Management Study
Acronym: MHM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Society for Vascular Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMRIMHM2018
Record Dates: First submitted 2018-02-02; First posted 2018-03-06 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Hypertension
Keywords: Hypertension; Telemonitoring; Digital Health
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: two randomized parallel groups. one group with standard care and one group with telemonitoring of blood pressure and hypertension.
Who Masked: Outcomes Assessor
Masking Description: the Data analysis will be performed by an independent team with masking the patients groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): This group is the usual standard treatment group
- Telemonitoring group (Other): This group will followed up with telemonitoring
  Interventions: Other: telemonitoring

INTERVENTIONS:
Other: telemonitoring — the follow-up of the patient will be performed with Telemonitoring
  Arms: Telemonitoring group

SUMMARY:
The present prospective study aims to assess the efficacy of using the telehealth solution "Hypertension Monitor" in patients with hypertension by comparison to the standard care.

DETAILED DESCRIPTION:
Although, meta-analysis confirms that BP telemonitoring may represent a useful tool to improve hypertension management, the strength of the provided evidence is limited. Therefore, future well-designed, large-sample, prospective, controlled trials are mandatory to understand the benefit of BP telemonitoring.

Recently, a specific telehealth solution for hypertension management has been developed in France (Hypertension Monitor - e-CoreLab®).

The present prospective study aims to assess the efficacy of using the telehealth solution "Hypertension Monitor" in patients with hypertension by comparison to the standard care.

The primary objective: To evaluate whether a home telehealth system can improve BP control and other risk factors in hypertensive individuals, as compared to the standard care.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Age between 18 and 80 years
* Patients with essential moderate Hypertension
* untreated or not adequately treated (need for treatment changes)
* Given written informed consent

Exclusion Criteria:

* Severe Hypertension (>180/110 mmHg)
* Difficulties to perform home blood pressure measurements
* Patients with arm circumference > 42 cm
* Night shift workers
* Body mass index > 35 kg/m²
* Atrial fibrillation and/or another arrhythmia
* Pregnancy
* Cardiovascular events (stroke, Myocardial infarction) in the last 6 months
* Severe Sleep Apnea Syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-06-03 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure (measured in clinic) | Primary objective after 3 month
  Systolic blood pressure will be measured in clinic according to the guidelines of the European Society of Hypertension (ESH).

SECONDARY OUTCOMES:
Timing to reach the blood pressure target | Evaluation performed at Month1 and Month 3
  how long we need to reach the Blood pressure normalization

CONTACTS AND LOCATIONS:
Overall Officials: ROLAND ASMAR, MD, Study Chair — Foundation-Medical research Institutes
Locations (1):
- Roland Asmar, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
the essential documents and the study results will be shared with all the investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study documents: Q1 2018 Study Results: Q2 2019
Access Criteria: the request will be reviewed by the scientific committee. Requestors will be required to sign an access agreement
URL: https://e-corelab.com/